CLINICAL TRIAL: NCT06010134
Title: Efficacy of Whole Body Vibration on Balance and Motor Control in Children With Osteogenesis Imperfecta
Brief Title: Osteogenesis Imperfecta and Balance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Nehad Ahmed Youness Abo-zaid, Assistant Professor of Pediatric Physical Therapy, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002577
Record Dates: First submitted 2023-08-17; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-05

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Whole Body Vibration; Balance; Motor Control
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Intervention Model Description: G 1 (control) received traditional physical therapy program for 30 min. G 2 (study) received traditional physical therapy program for 15 min. and Whole Body Vibration for 15 min
Who Masked: Participant
Masking Description: Double (Participant, Investigator) Single (Outcomes Assessor) Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group 1 (control group) and Group 2 (Whole Body Vibration group).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Group 1 the control group received selected physical therapy program which contain strengthening exercises for upper limb and lower limb muscles, stretching exercises for elbow extensors, hand pronator, wrist extensors, knee extensors and ankle dorsiflexors, coordination and balancing exercises.
  Interventions: Other: Physical Therapy Program
- Study group (Experimental): Group 2 the study group received the same physical therapy program 15 min. plus Whole Body Vibration for 15 min.
  Interventions: Other: Physical Therapy Program

INTERVENTIONS:
Other: Physical Therapy Program — Physical Therapy Program plus Whole Body Vibration

SUMMARY:
Osteogenesis Imperfecta (OI), also known as brittle bone disease, is a group of genetic disorders that mainly affect the bones. It results in bones that break easily. Its severity may be mild to severe. Other symptoms may include a blue tinge to the whites of the eye, short height, loose joints, hearing loss, breathing problems and problems with the teeth.

Physiotherapy is aimed to strengthen muscles and improve motility in a gentle manner, while minimizing the risk of fracture, and the use of support cushions to improve posture.

DETAILED DESCRIPTION:
This study aimed to assess the efficacy of Whole Body Vibration on balance and motor function in children with Osteogenesis Imperfecta.

Whole body vibration (WBV) therapy is targeted at musculoskeletal strengthening and has been trialed in a variety of conditions. WBV has been shown to have therapeutic advantage in various osteopenic preclinical models and populations such as postmenopausal women (improved mobility, muscle strength, postural strength, and bone density) and children with osteogenesis imperfecta (improved mobility)

ELIGIBILITY:
Inclusion Criteria:

1. Their age was ranging from six to twelve years
2. Children participated in this study were from both sexes
3. All children with stable medical and psychological status.
4. They were able to follow the verbal commands or instructions during testing.

Exclusion Criteria:

1. Children with visual or auditory problems.
2. Children with any cognitive problems.
3. Children without deformity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Over All Stabiity Index | at day 0
  Stability Index
Over All Stabiity Index | at day 90
  Stability Index
Medio lateral Stabiity Index | at day 0
  Stability Index
Medio lateral Stabiity Index | at day 90
  Stability Index
Antro posterior Stabiity Index | at day 0
  Stabiity Index
Antro posterior Stabiity Index | at day 90
  Stabiity Index

CONTACTS AND LOCATIONS:
Overall Officials: Hanady Mohamed, Principal Investigator — Faculty of Physical Therapy, Benha University
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andersen PE Jr, Hauge M. Osteogenesis imperfecta: a genetic, radiological, and epidemiological study. Clin Genet. 1989 Oct;36(4):250-5. doi: 10.1111/j.1399-0004.1989.tb03198.x. PMID 2805382
- [Result] Folkestad L, Hald JD, Ersboll AK, Gram J, Hermann AP, Langdahl B, Abrahamsen B, Brixen K. Fracture Rates and Fracture Sites in Patients With Osteogenesis Imperfecta: A Nationwide Register-Based Cohort Study. J Bone Miner Res. 2017 Jan;32(1):125-134. doi: 10.1002/jbmr.2920. Epub 2016 Aug 29. PMID 27448250
- [Result] Bishop N. Bone Material Properties in Osteogenesis Imperfecta. J Bone Miner Res. 2016 Apr;31(4):699-708. doi: 10.1002/jbmr.2835. Epub 2016 Mar 26. PMID 26987995
- [Result] Rauch F, Travers R, Parfitt AM, Glorieux FH. Static and dynamic bone histomorphometry in children with osteogenesis imperfecta. Bone. 2000 Jun;26(6):581-9. doi: 10.1016/s8756-3282(00)00269-6. PMID 10831929